CLINICAL TRIAL: NCT07044713
Title: A Comparison of the Use of Hand Puppets and Image Watching and Coloring Books for Children in Reducing Pain and Fear During Blood Collection Procedures
Brief Title: Use of Hand Puppets and Image Watching and Coloring Books for Children in During Blood Collection Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Gamze Akay, Assistant Professor, Artvin Coruh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hand Puppets, Image Watching
Record Dates: First submitted 2025-06-24; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Blood Collection
Keywords: blood collection; fear; child; pain; hand puppet; Tracing and Painting the Image
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Routine clinical care will be applied to the control group. No action will be taken.
- Experimental Group (Experimental): Before blood collection, the child will be shown games with hand puppets and will be asked to watch the image and color with the Coloring Book.
  Interventions: Other: Hand Puppet; Other: The Visual Viewing and Coloring Book

INTERVENTIONS:
Other: Hand Puppet — Children who come to the hospital's blood collection unit and meet the research criteria will be randomly assigned to the hand puppet group. The scales will be filled out by the nurse and the child five minutes before the blood collection. The researcher will benefit from the experiences of the child development specialist and preschool teacher before the research on puppet scenarios. In the interview room outside the blood collection unit, the child's parent will be asked to tell the researcher about the things the child enjoys and likes. The researcher will show the child puppet characters on various themes and the child will be asked to choose the puppet character he/she wants before the blood collection. The puppet scenarios will be improvised in light of the information received from the child's mother and father during the demonstration and will be shaped according to the child's wishes. In this way, the child will turn the scary hospital environment into an entertaining environm
  Arms: Experimental Group
Other: The Visual Viewing and Coloring Book — Children who come to the hospital's blood collection unit and meet the research criteria will be randomly assigned to the coloring group. The scales will be filled out by the nurse and the child five minutes before the blood is drawn. The Visual Viewing and Coloring Book consists of pictures that require coloring. The children will be given a book before the blood is drawn and will be asked to draw or color a picture as they prefer during the procedure. The fear scale will be assessed by the nurse and the child five minutes before, during, and five minutes after the procedure. The pain scale will be assessed by the nurse and the child during and five minutes after the procedure. The child will be shown the facial expressions on both the fear scale and the pain scale and asked which one it is, and the score corresponding to the facial expression he/she indicates will be recorded. Mothers will stay with their children during the treatment proce
  Arms: Experimental Group

SUMMARY:
The aim of this study was to compare a hand puppet with image viewing and a coloring book for children in reducing children's pain and fear during blood collection.

DETAILED DESCRIPTION:
Ninety volunteer children aged 3-6 coming for blood collection will be randomly divided into three groups: hand puppet, viewing and painting the image, and control group. Children will be assessed before, during, and after the procedure. Pain related to blood collection will be assessed with the Wong-Baker Faces Pain Scale, and fear will be assessed with the Child Fear Scale. In addition, children's demographic data will be recorded in the Information Form.

ELIGIBILITY:
Inclusion Criteria:

* Being between 3-6 years old
* Taking blood samples at once
* No visual-auditory and speech disorders
* Being open to communication and
* Being accompanied by a parent.

Exclusion Criteria:

* Having a chronic disease
* Having a visual-auditory and speech disorder
* History of sedative, analgesic or narcotic substance use within 24 hours before admission
* Children whose parents do not agree to participate in the study.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient Identification Form | Baseline
  It is a form consisting of 7 questions in total, including the child's age, gender, previous hospital experience, if any, how many times the child has been hospitalized, whether the parents have prepared for the blood collection process beforehand, experience of having blood drawn in the last six months, and reactions to the blood collection process. It was prepared by researchers in accordance with the literature.
Wong Baker Face Pain Scale | Baseline and up to 4 weeks
  Children between the ages of three and eight can express many pain areas and their severity. In this study, the Wong-Baker Pain Inventory will be used in combination with the Visual Analog Scale, since face scales are more appropriate. The Wong Baker Face Pain Scale was developed by Donna Wong and Connie Moran Baker in 1981. The scale is suitable for children between the ages of three and eighteen. The scale includes facial expressions that the child can enjoy and enjoy. For this reason, it has been stated that it gives more accurate results. The scale has scores of "0", "2", "4", "6", "8", and "10". A score of "0" indicates no pain and a score of "10" indicates the highest pain. This scale does not have a Cronbach's alpha score. It has been reported that reliability studies have not been conducted on such scales. In our study, the child will be shown the facial expressions on the pain scale and asked which one it is, and the score co
Child Fear Scale | Baseline and up to 4 weeks
  The Turkish validity of this scale, developed by McMurtry and colleagues, was done by Gerçeker and colleagues. The changes in the facial muscles of the frightened expression were drawn by a graphic artist from a photograph of a frightened face. It can be used by the parent, child or researcher to scale the child's fear. The scale, which has facial expressions scored from 0 to 4, is shown to the child. A score of 4 indicates that the child is very frightened, and a score of 0 indicates that the child is not frightened. It is accepted that a score of "0" indicates a neutral expression (no fear), a score of "1" indicates a very low level of fear, a score of "2" indicates a little fear, a score of "3" indicates a greater level of fear, and a score of 4 indicates that the level of fear is at the highest level. This scale can be used to measure fear before and during the procedure. In our study, the child will be shown the facial expressions on the

CONTACTS AND LOCATIONS:
Overall Officials: Gamze AKAY, 1, Principal Investigator — Artvin Coruh University
Locations (1):
- Kilis Prof. Dr. Alaeddin Yavaşca State Hospital, Kilis, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oluc T, Sarialioglu A. The effect of a hand puppet-based therapeutic play for preschool children on the fear and pain associated with blood collection procedure. J Pediatr Nurs. 2023 Sep-Oct;72:e80-e86. doi: 10.1016/j.pedn.2023.06.012. Epub 2023 Jun 15. PMID 37330277
- See also: Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/37330277/